CLINICAL TRIAL: NCT01963208
Title: A Multicenter, Double Blind, Randomized, Placebo-Controlled Trial to Determine the Efficacy and Safety of Ganaxolone as Adjunctive Therapy for Adults With Drug-Resistant Partial-Onset Seizures Followed by Long-term Open-Label Treatment
Brief Title: Phase 3 Study of Adjunctive Ganaxolone in Adults With Drug-resistant Partial Onset Seizures and Open-label Extension
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Marinus Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: 1042-0603
Record Dates: First submitted 2013-10-11; First posted 2013-10-16 (Estimated); Results first posted 2023-02-14 (Actual); Last update posted 2023-02-14 (Actual); Status verified 2023-01

CONDITIONS: Drug Resistant Partial Onset Seizure
Keywords: partial onset seizures; complex partial seizures; simple partial seizures; anticonvulsant; ganaxolone; neurosteroid; Marinus; epilepsy
MeSH Terms: conditions — Seizures; Epilepsies, Partial; Epilepsy | interventions — ganaxolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (6):
- Double Blind - Cohort 1 - Ganaxolone (Experimental): 1200 mg/day and 1800 mg/day + AED
  Interventions: Drug: ganaxolone
- Double Blind - Cohort 1 - Placebo (Placebo Comparator): Placebo + AED
  Interventions: Drug: Placebo
- Open Label - Ganaxolone in Double-blind phase (Experimental): 1800 mg/day + AED
  Interventions: Drug: ganaxolone
- Double Blind - Cohort 2 - Ganaxolone (Experimental): 1800 mg/day + AED
  Interventions: Drug: ganaxolone
- Double Blind - Cohort 2 - Placebo (Placebo Comparator): Placebo +AED
  Interventions: Drug: Placebo
- Open Label - Placebo in Double-blind phase (Experimental): 1800 mg/day + AED
  Interventions: Drug: ganaxolone

INTERVENTIONS:
Drug: ganaxolone — 200 mg and 225 mg capsules; target dose 1800 mg/day dosed 900mg 2x/day
  Other Names: gnx
  Arms: Double Blind - Cohort 1 - Ganaxolone; Double Blind - Cohort 2 - Ganaxolone; Open Label - Ganaxolone in Double-blind phase; Open Label - Placebo in Double-blind phase
Drug: Placebo — placebo
  Other Names: pbo
  Arms: Double Blind - Cohort 1 - Placebo; Double Blind - Cohort 2 - Placebo

SUMMARY:
The study will evaluate the effectiveness and safety of an investigational drug-ganaxolone - on partial seizure frequency in adults with epilepsy taking a maximum of 3 antiepileptic medications (AEDs).

DETAILED DESCRIPTION:
This is a 2-cohort study comprised of 2 phases in each cohort. Phase 1 is a double-blind (DB) phase followed by Phase 2, an open-label phase. Cohort 1 will provide tolerability, safety, and PK information for ganaxolone 1200 milligram per day (mg/day), 1800 mg/day and placebo. Cohort 2 will investigate the efficacy, tolerability and safety of ganaxolone 1800 mg/day compared to placebo. Cohort 1 (N= approximately 50) will enroll into a 67-week study comprised of a 4-week prospective baseline period plus 4 week retrospective baseline followed by two treatment phases: a 9-week randomized DB placebo-controlled treatment phase followed by a 52-week open label treatment phase. Cohort 2 (N=150) will enroll into a 72-week study comprised of a 8-week prospective baseline period followed by two treatment phases: a 14-week randomized DB placebo-controlled treatment phase followed by a 52-week open label treatment phase.

ELIGIBILITY:
Inclusion Criteria:

* Able to give informed consent in writing, or have a legally authorized representative able to do so
* Willing to enter and participate for the full term of the double blind phase and willing to enter into the open-label phase
* Male or female outpatients > 18 years of age
* Have a confident diagnosis of drug-resistant epilepsy with partial-onset seizures (POS), with or without secondary generalization, for ≥2 years. Have residual POS despite having been treated in the past with at least 2 approved anti-epilepsy drugs (AEDs) either alone or in combination
* Based on history, participants would be anticipated to have at least 3 POS during each 4-week Baseline period and unlikely to have 21 or more consecutive POS-free days
* Currently being treated and maintained with a stable regimen of 1, 2, or 3 AEDs
* Able and willing to maintain daily seizure calendar
* Able and willing to take drug with food twice daily
* Sexually active women of childbearing potential must use acceptable birth control and have a negative pregnancy test at all visits

Exclusion Criteria:

* Have had previous exposure to ganaxolone
* Known sensitivity or allergy to any component in the study drug, progesterone, or other related steroid compounds
* Exposure to any investigational drug or device <30 days prior to screening, or plans to take another investigational drug at any time during the study
* Time of onset of epilepsy treatment <2 years prior to enrollment
* Have generalized epilepsy, such as Lennox-Gastaut syndrome, juvenile myoclonic epilepsy, absence epilepsy, or non-epileptic seizures within the last 12- month period prior to study entry
* Have less than 3 POS seizures in a 28-day period or more than 21 consecutive seizure-free days during the Baseline period
* Have only simple partial seizures without any observable motor component
* Have innumerable seizures or status epilepticus within the last 12-months prior to screening
* Have more than 100 POS per 4-week Baseline period
* Have seizures secondary to illicit drug or alcohol use, infection, neoplasm, demyelinating disease, degenerative neurological disease, or central nervous system (CNS) disease deemed progressive, metabolic illness, or progressive degenerative disease
* Current use of vigabatrin is not permitted. If prior use of vigabatrin, must have documented stable visual fields
* Current use of ezogabine is not permitted. If prior use, must have been off the medication for at least 3 months prior to screening and have had documented normal fundoscopic exam by ophthalmologist
* Are planning surgery, or to be evaluated for surgery, during the double-blind phase to control seizures including VNS implantation
* Are suffering from acute or progressive neurological disease, moderate or severe psychiatric disease, or severe mental abnormalities that are likely to require changes in drug therapy during the double-blind portion of the study or interfere with the objectives of the study or the ability to adhere to the protocol requirements
* Have a history of an actual suicide attempt in the last 5 years or more than 1 lifetime suicide attempt
* Have a positive urine drug screen at Screening or meet criteria for current or historical Substance Use Disorder (DSM-V criteria) within the past 5 years.
* Have any medical condition that, in the investigator's judgment, is considered to be clinically significant and could potentially affect participant safety or study outcome, including but not limited to: clinically significant cardiac, renal, pulmonary, gastrointestinal, hematologic or hepatic conditions; or a condition that affects the absorption, distribution, metabolism or excretion of drugs
* Have elevated ALT (SGPT) or AST (SGOT) greater than 3 times upper limits of normal, or total bilirubin greater than 1.5 times ULN
* Have a history of malignancy within the past 2 years, with the exception of basal cell carcinoma
* Are currently following or planning to follow a ketogenic diet
* Use of dietary supplements or herbal preparations are not permitted if participant has been using them consistently for less than 6 months prior to screening, or does not plan on remaining on stable doses for the duration of the double blind phase. Use of St. John's Wort is not permitted
* Females who are pregnant, currently breastfeeding or planning to become pregnant during the duration of the study
* A history of chronic noncompliance with drug regimens
* Inability to withhold grapefruit and grapefruit juice from diet during the entire clinical trial

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 405 (Actual)
Dates: Start 2013-10; Primary Completion 2016-05 (Actual); Study Completion 2016-10 (Actual)

CONTACTS AND LOCATIONS:
Locations (68):
- United States (33):
  - University of Alabama Epilepsy Center, Birmingham, Alabama
  - University of Alabama at Birmingham, Birmingham, Alabama
  - Xenoscience Inc., Phoenix, Arizona
  - The MORE Foundation, Sun City, Arizona
  - Clinical Trials Inc., Little Rock, Arkansas
  - Neuro-Pain Medical Center, Inc, Fresno, California
  - Neurological Research Institute, Santa Monica, California
  - University of Colorado- Anschutz Outpatient Pavilion, Aurora, Colorado
  - Neuroscience Consulants, Miami, Florida
  - Medsol Clinical Research Center, Port Charlotte, Florida
  - Consultants in Epilepsy & Neurology, Boise, Idaho
  - Bluegrass Epilepsy Research, LLC, Lexington, Kentucky
  - Mid-Atlantic Epilepsy Center, Bethesda, Maryland
  - Bringham and Women's Hospital, Boston, Massachusetts
  - Minneapolis Clinic of Neurology, Golden Valley, Minnesota
  - The Comprehensive Epilepsy Care Center for Children and Adults, Chesterfield, Missouri
  - Cooper Medical Center of Rowan University, Camden, New Jersey
  - Northeast Regional Epilepsy Group, Hackensack, New Jersey
  - Five Towns Neuroscience Research, Cedarhurst, New York
  - Northeast Regional Epilepsy Group, Middletown, New York
  - Winthrop University Hospital, Mineola, New York
  - New York University Comprehensive Epilepsy Center, New York, New York
  - Northeast Regional Epilepsy Group, New York, New York
  - Wake Forest Health Sciences, Winston-Salem, North Carolina
  - Ohio Clinical Research Partners, LLC, Canton, Ohio
  - Ohio State University, Columbus, Ohio
  - Lynn Health Institute, Oklahoma City, Oklahoma
  - Sooner Clinical Research, Oklahoma City, Oklahoma
  - Jefferson Comprehensive Epilepsy Center, Philadelphia, Pennsylvania
  - Temple University School of Medicine, Philadelphia, Pennsylvania
  - Neurology Consultants of Dallas, Dallas, Texas
  - Texas Epilepsy Group, Dallas, Texas
  - Rainier Clinical Research Center, Inc., Renton, Washington
- Australia (7):
  - Royal Prince Alfred Hospital, Camperdown, New South Wales
  - The Prince of Wales Hospital, Randwick, New South Wales
  - Westmead Hospital, Westmead, New South Wales
  - Flinders Medical Center, Bedford Park, South Australia
  - St. Vincent's Hospital, Fitzroy, Victoria
  - The Florey Institute of Neuroscience and Mental Health, Heidelberg, Victoria
  - The Royal Melbourne Hospital, Parkville, Victoria
- Bulgaria (8):
  - MHAT, Blagoevgrad
  - UMHAT Dr. Georgi Stranski Clinic of Neurology, Pleven
  - Medical Centre-Teodora, Rousse
  - Medical Center Excelsior 4, Sofia
  - SHATNP, Sofia
  - MHAT Lyulin Department of Neurology, Sofia
  - UMHAT Alexandrovska Clinic of Nerve Diseases, Sofia
  - Medical Center Ekvita Ltd, Varna
- Germany (6):
  - Epilepsieklinik, Bernau
  - Krankenhaus Mara Epilepsie-Zentrum, Bielefeld
  - Klinik fur Epileptologie, Bonn
  - Neuro-Consil, Dussseldorf
  - Universitatsklinikum GieBen und Marburg, Marburg
  - Universitatsklin Kum Ulm, Ulm
- Poland (6):
  - Novo-Med, Jaworowa
  - Centrum Medycne Dendryt, Katowice
  - Indywidualna Praktyka ul Narutowicza, Lublin
  - Wojewodzki Szpital Specjalistyczny Oddzial, Lublin
  - Fundacja Epileptologii Wiertnicza, Warsaw
  - Instytut Psychiatrii i Neurologii, Warsaw
- Russia (8):
  - Kazan State Medical University, Kazan'
  - Moscow
  - Nizhny Novgorod
  - Novosibirsk
  - City Neurological Center, Novosibirsk
  - Saint Petersburg
  - Samara
  - Yaroslavl

RESULTS

PARTICIPANT FLOW:
Recruitment Details: This was a 2-cohort study where each cohort comprised of 2 treatment phases. Phase 1 was a double-blind phase followed by Phase 2, an open-label phase. The study analyzed safety, tolerability and pharmacokinetics (PK) of Ganaxolone when compared with placebo in both the cohorts.
Pre-assignment Details: A total of 405 participants were enrolled in the study. Double Blind: Cohort 1 comprised of Titration period (Week 0 to Week 1) and Maintenance period (Week 1 to Week 9). Double Blind: Cohort 2 comprised of Titration period (Week 0 to Week 2) and Maintenance period (Week 2 to Week 14).
Groups:
- Double Blind: Cohort 1 - Ganaxolone: Participants were administered ganaxolone 1200 milligrams per day (mg/day) and 1800 mg/day + Antiepileptic drug (AED). Following the completion of the double-blind phase, participants randomized to placebo were transitioned to ganaxolone while participants randomized to ganaxolone remained on the drug at 1800 mg/day in the open-label phase.
- Double Blind: Cohort 1 - Placebo; Double Blind: Cohort 2 - Placebo: Participants were administered Placebo + AED. Following the completion of the double-blind phase, participants randomized to placebo were transitioned to ganaxolone while participants randomized to ganaxolone remained on the drug at 1800 mg/day in the open-label phase.
- Double Blind: Cohort 2 - Ganaxolone: Participants were administered Ganaxolone 1800 mg/day + AED. Following the completion of the double-blind phase, participants randomized to placebo were transitioned to ganaxolone while participants randomized to ganaxolone remained on the drug at 1800 mg/day in the open-label phase.
- Open Label: Ganaxolone in Double-blind Phase: Following the completion of the double-blind phase, participants randomized to ganaxolone remained on the drug at 1800 mg/day + AED. Participants from Double Blind: Cohort 1 - Ganaxolone and Double Blind: Cohort 2 - Ganaxolone were combined to enter in Open Label: Ganaxolone in Double-blind Phase
- Open Label: Placebo in Double-blind Phase: Following the completion of the double-blind phase, participants randomized to placebo were transitioned to ganaxolone + AED. Participants from Double Blind: Cohort 1 - Placebo and Double Blind: Cohort 2 - Placebo were combined to enter in Open Label: Placebo in Double-blind Phase
Period: Treatment Phase 1 (Up to Week 14)
Arm/Group | Double Blind: Cohort 1 - Ganaxolone | Double Blind: Cohort 1 - Placebo | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo | Open Label: Ganaxolone in Double-blind Phase | Open Label: Placebo in Double-blind Phase
Started | 24 | 22 | 179 | 180 | 0 | 0
Completed | 23 | 19 | 135 | 154 | 0 | 0
Not Completed | 1 | 3 | 44 | 26 | 0 | 0
Not completed — Adverse Event | 1 | 0 | 30 | 11 | 0 | 0
Not completed — Withdrawal by Subject | 0 | 2 | 8 | 9 | 0 | 0
Not completed — Non-compliance | 0 | 0 | 4 | 0 | 0 | 0
Not completed — Protocol Violation | 0 | 0 | 1 | 3 | 0 | 0
Not completed — Other | 0 | 1 | 1 | 1 | 0 | 0
Not completed — Insufficient Clinical Response | 0 | 0 | 0 | 1 | 0 | 0
Not completed — Lost to Follow-up | 0 | 0 | 0 | 1 | 0 | 0
Period: Treatment Phase 2 (Up to Week 68)
Arm/Group | Double Blind: Cohort 1 - Ganaxolone | Double Blind: Cohort 1 - Placebo | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo | Open Label: Ganaxolone in Double-blind Phase | Open Label: Placebo in Double-blind Phase
Started | 0 | 0 | 0 | 0 | 158 | 173
Completed | 0 | 0 | 0 | 0 | 57 | 44
Not Completed | 0 | 0 | 0 | 0 | 101 | 129
Not completed — Adverse Event | 0 | 0 | 0 | 0 | 16 | 15
Not completed — Withdrawal by Subject | 0 | 0 | 0 | 0 | 7 | 19
Not completed — Non-Compliance | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Protocol Violation | 0 | 0 | 0 | 0 | 0 | 1
Not completed — Other | 0 | 0 | 0 | 0 | 58 | 75
Not completed — Insufficient Clinical Response | 0 | 0 | 0 | 0 | 20 | 17
Not completed — Death | 0 | 0 | 0 | 0 | 0 | 1

BASELINE CHARACTERISTICS:
Population: Modified intent to treat (mITT) population: all randomized participants who received at least 1 dose of study medication and provided any post Baseline seizure outcome data.
Groups:
- Double Blind: Cohort 1 - Ganaxolone: Participants were administered ganaxolone 1200 mg/day and 1800 mg/day + AED. Following the completion of the double-blind phase, participants randomized to placebo were transitioned to ganaxolone while participants randomized to ganaxolone remained on the drug at 1800 mg/day in the open-label phase.
- Total: Total of all reporting groups
Arm/Group | Double Blind: Cohort 1 - Ganaxolone | Double Blind: Cohort 1 - Placebo | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo | Total
Number analyzed (Participants) | 24 | 21 | 178 | 172 | 395
Age, Continuous [Mean (Standard Deviation); unit: Years] | 35.1 (10.25) | 41.1 (11.83) | 40.6 (12.48) | 42.1 (12.37) | 39.72 (11.73)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 13 | 12 | 113 | 97 | 235
  Male | 11 | 9 | 65 | 75 | 160
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 2 | 2 | 11 | 11 | 26
  Not Hispanic or Latino | 22 | 19 | 167 | 161 | 369
  Unknown or Not Reported | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 1 | 1
  Asian | 0 | 1 | 3 | 3 | 7
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
  Black or African American | 1 | 0 | 3 | 4 | 8
  White | 22 | 19 | 167 | 160 | 368
  More than one race | 0 | 0 | 0 | 0 | 0
  Unknown or Not Reported | 1 | 1 | 5 | 4 | 11

OUTCOME MEASURES:

1. Primary Outcome: Double Blind: Cohort 2: Percent Change From Baseline in 28-day Seizure Frequency During Titration + Maintenance Period
Description: Seizure frequency was based on the number of seizures per 28 days, calculated as the number of seizures over the time interval multiplied by 28 and divided by the number of days in the interval. Baseline 28-day seizure frequency was calculated as the number of seizures in the Baseline period (≤ 56 days) divided by the number of days with available seizure data in the Baseline period and multiplied by 28. Baseline was defined as non-missing value of last assessment before first dose. Primary analysis was performed using a rank analysis of covariance (ANCOVA).
Time Frame: Baseline and Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 178 | 172
Percent change | -21.28 [-29.60 to -14.29] | -10.25 [-20.14 to -1.28]
Statistical Analysis 1: Comparison: Double Blind: Cohort 2 - Ganaxolone vs Double Blind: Cohort 2 - Placebo; Test type: Other; p = 0.1788, Rank ANCOVA — The null hypothesis is that there is no difference between the distributions of the two treatment groups with respect to percent change in seizure frequency; Median Difference (Final Values) = -7.06, 95% CI 2-sided [-17.44 to 3.52]

2. Secondary Outcome: Double Blind: Cohort 2: Number of Participants With ≥50% Responder Rate During Titration + Maintenance Period
Description: A 50% responder was a participant who experienced at least a 50% decrease in 28-day seizure frequency compared to Baseline.
Time Frame: Up to Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 178 | 172
Participants | 50 | 39

3. Secondary Outcome: Double Blind: Cohort 2: Change From Baseline in the Number of Seizure Free Days Per 28-day Period During Titration + Maintenance Period
Description: Baseline number of seizure free days per 28-day period was calculated as: the number of seizure free days in the entire Baseline period (<=56 days) divided by the number of days with available seizure data in the baseline period and multiplied by 28. Post-Baseline number of seizure free days per 28-day period was calculated as: the number of seizure free days in the entire treatment period divided by the number of days with available seizure data in the treatment period and multiplied by 28. Change from Baseline in number of seizure free days per 28-day period from Baseline was calculated as: Post-Baseline number of seizure free days per 28-day period minus Baseline number of seizure free days per 28-day period. Baseline was defined as non-missing value of last assessment before first dose.
Time Frame: Baseline and Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Seizure free days
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 178 | 172
Seizure free days | 1.47 (4.396) | 1.01 (4.223)

4. Secondary Outcome: Double Blind: Cohort 2: Number of Participants With Clinical Global Impression of Change - Improvement (CGI-I) at Week 14
Description: The CGI-I scale is a clinician-rated 7-point Likert scale used to assess the degree to which the participant's epilepsy symptoms have changed relative to Baseline. It was rated as 1. "very much improved"; 2. "much improved"; 3. "minimally improved"; 4. "no change"; 5. "minimally worse"; 6. "much worse"; 7. "very much worse". Higher scores indicated worse condition. Baseline was defined as non-missing value of last assessment before first dose.
Time Frame: At Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 140 | 159
Participants
  Very much improved | 7 | 5
  Much improved | 28 | 30
  Minimally improved | 41 | 47
  No change | 56 | 67
  Minimally worse | 6 | 8
  Much worse | 2 | 2
  Very much worse | 0 | 0

5. Secondary Outcome: Double Blind: Cohort 2: Percent Change From Baseline in 28-day Seizure Frequency During Maintenance Period
Description: Seizure frequency was based on the number of seizures per 28 days, calculated as the number of seizures over the time interval multiplied by 28 and divided by the number of days in the interval. Baseline 28-day seizure frequency was calculated as the number of seizures in the Baseline period (≤ 56 days) divided by the number of days with available seizure data in the Baseline period and multiplied by 28. Baseline was defined as non-missing value of last assessment before first dose.
Time Frame: Baseline and Week 2 to Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Median (95% Confidence Interval); unit: Percent change
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 166 | 169
Percent change | -20.56 [-31.56 to -12.69] | -12.50 [-20.78 to -3.03]

6. Secondary Outcome: Double Blind: Cohort 2: Change From Baseline in 28-day Seizure Frequency During Titration + Maintenance Period
Description: Seizure frequency was based on the number of seizures per 28 days, calculated as the number of seizures over the time interval multiplied by 28 and divided by the number of days in the interval. Baseline 28-day seizure frequency was calculated as the number of seizures in the Baseline period (≤ 56 days) divided by the number of days with available seizure data in the Baseline period and multiplied by 28. Baseline was defined as non-missing value of last assessment before first dose. Change from Baseline was calculated by subtracting Baseline value from the post-dose visit value.
Time Frame: Baseline and Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Seizures per 28 days
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 178 | 172
Seizures per 28 days | -1.46 (9.650) | -0.33 (11.040)

7. Secondary Outcome: Double Blind: Cohort 2: Change From Baseline in 28-day Seizure Frequency During Maintenance Period
Description: as for outcome 6
Time Frame: Baseline and Week 2 to Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Seizures per 28 days
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 166 | 169
Seizures per 28 days | -1.67 (11.809) | -0.64 (12.153)

8. Secondary Outcome: Double Blind: Cohort 2: Change From Baseline in the Number of Seizure Free Days Per 28-day Period During Maintenance Period
Description: Baseline number of seizure free days per 28-day period was calculated as: the number of seizure free days in the entire Baseline period (≤ 56 days) divided by the number of days with available seizure data in the Baseline period and multiplied by 28. Post-Baseline number of seizure free days per 28-day period was calculated as: the number of seizure free days in the entire treatment period divided by the number of days with available seizure data in the treatment period and multiplied by 28. Change from Baseline in number of seizure free days per 28-day period from Baseline was calculated as: Post-Baseline number of seizure free days per 28-day period minus Baseline number of seizure free days per 28-day period. Baseline was defined as non-missing value of last assessment before first dose.
Time Frame: Baseline and Week 2 to Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Seizure free days
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 166 | 169
Seizure free days | 1.63 (4.824) | 1.20 (4.462)

9. Secondary Outcome: Double Blind: Cohort 2: Percentage of Responders Experiencing a ≥R% (80%, 60%, 40%, and 20%) Reduction From Baseline to the End of Treatment Period in 28-day Seizure Frequency During Titration + Maintenance Period
Description: Percentage of participants who had reductions of ≥ 80%, ≥ 60%, ≥ 40%, and ≥ 20% in 28-day seizure frequency from Baseline is presented. A responder is an individual whose reduction of percent change from Baseline in 28-day seizure frequency was ≥ 50%. Baseline was defined as non-missing value of last assessment before first dose.
Time Frame: Up to Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 178 | 172
Percentage of participants
  Reduction ≥ 80% | 7.3 | 2.33
  Reduction ≥ 60% | 20.79 | 16.86
  Reduction ≥ 40% | 33.15 | 29.65
  Reduction ≥ 20% | 51.69 | 43.6

10. Secondary Outcome: Double Blind: Cohort 2: Percentage of Responders Experiencing a ≥R% (80%, 60%, 40%, and 20%) Reduction From Baseline to the End of Treatment Period in 28-day Seizure Frequency During Maintenance Period
Description: as for outcome 9
Time Frame: Week 2 to Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 178 | 172
Percentage of participants
  Reduction ≥ 80% | 8.43 | 5.81
  Reduction ≥ 60% | 24.16 | 18.02
  Reduction ≥ 40% | 33.71 | 31.4
  Reduction ≥ 20% | 47.19 | 42.44

11. Secondary Outcome: Double Blind: Cohort 2: Percentage of Seizure Free Participants During the Maintenance Period
Description: Percentage of participants who completed the study without any seizures is presented
Time Frame: Week 2 to Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 178 | 172
Percentage of participants | 1.12 | 0

12. Secondary Outcome: Double Blind: Cohort 2: Percentage of Participants Who Experienced at Least One 28-day Seizure Free Period During Titration + Maintenance Phase
Description: Percentage of participants who experienced at least one 28-day seizure free period is presented
Time Frame: Up to Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Number; unit: Percentage of participants
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 178 | 172
Percentage of participants | 17.98 | 18.02

13. Secondary Outcome: Double Blind: Cohort 2: Longest Percent of Time Spent Seizure-free During Titration + Maintenance Period
Description: The longest period of time seizure-free was defined as the percent of the longest seizure-free period (days) divided by the days with available seizure data, and then multiplied by 100%.
Time Frame: Up to Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percentage of time spent
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 178 | 172
Percentage of time spent | 24.00 (22.457) | 17.58 (12.743)

14. Secondary Outcome: Double Blind: Cohort 2: Percent Change From Baseline in 28-day Seizure Frequency for Different Subtypes of Seizures During Titration + Maintenance Period
Description: Seizure frequency was based on the number of seizures per 28 days, calculated as the number of seizures over the time interval multiplied by 28 and divided by the number of days in the interval. The analysis was conducted for Partial-Onset Seizure (POS) only which included seizure subtypes: Complex partial seizures (CPS), secondarily generalized tonic-clonic (SGTC) seizures, simple partial seizure with motor/observable component (SPS-Motor) and Simple partial seizure (SPS) without motor/observable component. Baseline 28-day seizure frequency was calculated as the number of seizures in the Baseline period (≤ 56 days) divided by the number of days with available seizure data in the Baseline period and multiplied by 28. Baseline was defined as non-missing value of last assessment before first dose.
Time Frame: Baseline and Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Mean (Standard Deviation); unit: Percent change
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 150 | 152
Percent change
  CPS | -4.70 (92.373) | -6.52 (59.126)
  SGTC: number analyzed (Participants) | 69 | 82
  SGTC | -27.42 (69.394) | 1.02 (118.444)
  SPS-Motor: number analyzed (Participants) | 44 | 32
  SPS-Motor | -5.52 (93.228) | -21.97 (52.473)
  SPS: number analyzed (Participants) | 33 | 31
  SPS | 12.57 (129.979) | -3.53 (87.071)

15. Secondary Outcome: Double Blind: Cohort 2: Number of Participants With Patient Global Impression of Change - Improvement (PGI-I) at Week 8 and Week 14
Description: The PGI-I scale was a 7-point Likert scale completed by the Patient or Caregiver representing the degree to which the participant's epilepsy symptoms had changed relative to Baseline. It was rated as 1. "very much improved"; 2. "much improved"; 3. "minimally improved"; 4. "no change"; 5. "minimally worse"; 6. "much worse"; 7. "very much worse". Higher score indicated worse condition. Baseline was defined as non-missing value of last assessment before first dose.
Time Frame: Week 8 and Week 14
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 166 | 161
Participants
  Week 8: Very Much Improved | 7 | 5
  Week 8: Much Improved | 30 | 21
  Week 8: Minimally Improved | 44 | 51
  Week 8: No Change | 59 | 65
  Week 8: Minimally Worse | 12 | 11
  Week 8: Much Worse | 8 | 4
  Week 8: Very Much Worse | 6 | 4
  Week 14: Very Much Improved | 7 | 10
  Week 14: Much Improved | 33 | 29
  Week 14: Minimally Improved | 43 | 43
  Week 14: No Change | 46 | 60
  Week 14: Minimally Worse | 7 | 12
  Week 14: Much Worse | 3 | 4
  Week 14: Very Much Worse | 1 | 1

16. Secondary Outcome: Double Blind: Cohort 2: Number of Participants With Clinical Global Impression of Change - Improvement (CGI-I) at Week 8
Description: as for outcome 4
Time Frame: At Week 8
Population: mITT Population. Only those participants with data available at the specified data points were analyzed.
Measure: Count of Participants; unit: Participants
Arm/Group | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo
Number analyzed (Participants) | 166 | 162
Participants
  Very much improved | 3 | 4
  Much improved | 27 | 20
  Minimally improved | 50 | 49
  No change | 68 | 71
  Minimally worse | 8 | 12
  Much worse | 9 | 5
  Very much worse | 1 | 1

ADVERSE EVENTS:
Time Frame: Week -8 through Week 14 in Double blind phase and from Week 16 to Week 68 in open label phase
Description: Safety Population: included all randomized participants who received at least 1 dose of study medication.
Arm/Group | Double Blind: Cohort 1 - Ganaxolone | Double Blind: Cohort 1 - Placebo | Double Blind: Cohort 2 - Ganaxolone | Double Blind: Cohort 2 - Placebo | Open Label: Ganaxolone in Double-blind Phase | Open Label: Placebo in Double-blind Phase
All-Cause Mortality (participants affected / at risk) | 0/24 | 0/21 | 0/179 | 0/176 | 0/158 | 1/173
Serious Adverse Events (participants affected / at risk) | 0/24 | 0/21 | 9/179 | 9/176 | 12/158 | 12/173
Other Adverse Events (participants affected / at risk) | 10/24 | 3/21 | 91/179 | 42/176 | 42/158 | 67/173
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind: Cohort 1 - Ganaxolone (N=24) | Double Blind: Cohort 1 - Placebo (N=21) | Double Blind: Cohort 2 - Ganaxolone (N=179) | Double Blind: Cohort 2 - Placebo (N=176) | Open Label: Ganaxolone in Double-blind Phase (N=158) | Open Label: Placebo in Double-blind Phase (N=173)
Coronary artery disease (Cardiac disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Small intestinal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Oesophageal obstruction (Gastrointestinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Gait disturbance (General disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (2)
Asthenia (Gastrointestinal disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Pneumonia (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Lung abscess (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Pulmonary tuberculosis (Infections and infestations) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Meningitis viral (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Appendicitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Clostridium difficile colitis (Infections and infestations) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Tongue injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Foot fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Subdural haematoma (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Spinal column injury (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Fall (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Accidental overdose (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ankle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Clavicle fracture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Ligament rupture (Injury, poisoning and procedural complications) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Hypokalaemia (Metabolism and nutrition disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Rhabdomyolysis (Musculoskeletal and connective tissue disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 2 (2) | 2 (2) | 1 (1) | 4 (4)
Epilepsy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1)
Grand mal convulsion (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (2)
Seizure cluster (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Status epilepticus (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Toxic encephalopathy (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Hallucination (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Anxiety (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1)
Confusional state (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 1 (1)
Delusion (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1)
Depression (Psychiatric disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 0 (0)
Mental status changes (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Suicidal ideation (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 1 (1) | 0 (0)
Suicide attempt (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0)
Somnolence (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Speech disorder (Nervous system disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
Postictal psychosis (Nervous system disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Psychogenic seizure (Psychiatric disorders) | 0 (0) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0)
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 (0) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0)
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Double Blind: Cohort 1 - Ganaxolone (N=24) | Double Blind: Cohort 1 - Placebo (N=21) | Double Blind: Cohort 2 - Ganaxolone (N=179) | Double Blind: Cohort 2 - Placebo (N=176) | Open Label: Ganaxolone in Double-blind Phase (N=158) | Open Label: Placebo in Double-blind Phase (N=173)
Somnolence (Nervous system disorders) | 3 (3) | 2 (2) | 40 (50) | 8 (8) | 12 (13) | 29 (33)
Dizziness (Nervous system disorders) | 2 (3) | 0 (0) | 34 (44) | 9 (9) | 8 (16) | 27 (29)
Headache (Nervous system disorders) | 2 (2) | 0 (0) | 16 (17) | 15 (15) | 9 (15) | 11 (12)
Balance disorder (Nervous system disorders) | 2 (2) | 0 (0) | 5 (5) | 1 (1) | 3 (3) | 1 (1)
Ataxia (Nervous system disorders) | 3 (4) | 0 (0) | 3 (3) | 0 (0) | 2 (2) | 2 (3)
Dysarthria (Nervous system disorders) | 2 (2) | 0 (0) | 1 (1) | 1 (1) | 2 (2) | 4 (4)
Sedation (Nervous system disorders) | 3 (3) | 0 (0) | 1 (1) | 0 (0) | 1 (1) | 1 (2)
Nasopharyngitis (Infections and infestations) | 0 (0) | 0 (0) | 5 (5) | 9 (9) | 6 (6) | 9 (9)
Fatigue (General disorders) | 2 (2) | 0 (0) | 21 (28) | 12 (12) | 9 (10) | 15 (19)
Night sweats (General disorders) | 0 (0) | 1 (1) | 0 (0) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (2):
  • Study Protocol (2016-04-08): https://cdn.clinicaltrials.gov/large-docs/08/NCT01963208/Prot_000.pdf
  • Statistical Analysis Plan (2016-05-24): https://cdn.clinicaltrials.gov/large-docs/08/NCT01963208/SAP_001.pdf